CLINICAL TRIAL: NCT02355990
Title: Minimally Invasive Micro Sclerostomy First in Man Safety and Preliminary Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAN-FIM-1
Record Dates: First submitted 2015-01-31; First posted 2015-02-04 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Primary Open Angle Glaucoma; Pigmentary Glaucoma; Pseudoexfoliative Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIMS (Experimental): Minimally Invasive Micro Sclerostomy
  Interventions: Procedure: Minimally Invasive Micro Sclerostomy

INTERVENTIONS:
Procedure: Minimally Invasive Micro Sclerostomy — Creation of a drainage channel of 50 - 100 microns (diameter) at the sclera-corneal junction and extending from the anterior chamber to the interface between the sclera and the conjunctiva (subconjuctival space).

SUMMARY:
The study objective is to demonstrate the safety of Minimally Invasive Micro Sclerostomy (MIMS) device for lowering elevated IOP in patients diagnosed with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* End Stage primary open-angle glaucoma, pseudoexfoliation glaucoma or pigmentary glaucoma in the study eye (EGS criteria)
* Optic nerve appearance characteristic of glaucoma in the study eye
* Best-corrected visual acuity (BCVA) of counting-fingers, hand movements, light perception or no light perception due to glaucomatous loss of central vision in the study eye
* Patient is treated with 1 to 5 hypotensive medications in the study eye
* Unsatisfactory medicated IOP (≥ 18 mmHg) at the screening visit in the study eye
* Shaffer grade ≥ III in all four angle quadrants in the study eye
* Subject is able and willing to attend all scheduled follow-up exams
* Subject understands and signs the informed consent

Exclusion Criteria:

* Subjects presenting 1 or more of the following criteria will not be enrolled in the trial:

  * Ocular conditions with a poorer prognosis in the fellow eye than in the study eye
  * Closed angle forms of glaucoma in either eye
  * Congenital or developmental glaucoma in either eye
  * Other secondary glaucoma (such as neovascular, uveitic, lens-induced, trauma-induced, or glaucoma associated with increased episcleral venous pressure) in the study eye
  * Peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities in the study eye
  * Subject has history of penetrating keratoplasty (PKP)
  * Any previous surgery in the study eye (except for clear corneal cataract surgery) where the conjunctiva is not intact and elastic.
  * Any ocular disease or history in study eye such as severe dry eye, active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, and ocular pathology that may interfere with accurate IOP measurements
  * Prior surgery for an ab-interno or ab-externo device implanted in or through the Schlemm's canal in the study eye.
  * Use of oral hypotensive medication for glaucoma for treatment of the fellow eye
  * Less than the minimum visual function required for driving in the fellow eye: best-corrected visual acuity worse than 20/40 (Snellen equivalent) or Esterman visual field score less than 85%.
  * History of idiopathic or autoimmune uveitis in either eye
  * Severe trauma in study eye
  * active iris neovascularization, previous cyclodestructive procedure, prior scleral buckling procedure, presence of silicone oil, need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery in study eye within 12 month period
  * Vitreous present in anterior chamber, prior vitrectomy or virteous hemorrhage in study eye
  * Aphakia
  * Prior vitreoretinal surgery in study eye
  * Clinically significant ocular inflammation or infection within 90 days prior to screening
  * Unable to discontinue use of blood thinners in accordance with surgeon's standard preoperative instructions
  * Uncontrolled systemic disease that in the opinion of the investigator would put the subject's health at risk and/or prevent the subject from completing all study visits
  * Current participation or participation in another investigational drug or device clinical trial within the last 30 days before screening visit
  * Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Overall incidence of serious adverse events | 12 weeks

SECONDARY OUTCOMES:
Incidence of serious adverse events | 24 weeks
intraocular pressure (IOP) between 6 mmHg and 15 mmHg without medication | 24 weeks
Change in number of glaucoma medications from baseline in the study eye | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cotlear, MD, Principal Investigator
Locations (1):
- Goldschleger Eye Institute, The Chaim Sheba Medical Center, Tel Litwinsky, Israel